CLINICAL TRIAL: NCT00006194
Title: Effects of Exercise on Markers of Inflammation in Skeletal Muscle in Elderly Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0764; M01RR000036 (NIH)
Record Dates: First submitted 2000-09-07; First posted 2000-09-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Hip Fractures; Muscular Atrophy
Keywords: sarcopenia
MeSH Terms: conditions — Hip Fractures; Muscular Atrophy; Sarcopenia | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
Decreased skeletal muscle mass is a prevalent condition among the elderly, and an important cause of disability and functional decline. The declines in muscle mass associated with aging may be related to alterations in specific kinds of growth factors in the muscle. Elderly hip fracture patients often have significant decreases in muscle mass. The purpose of this study is to investigate whether an exercise program can induce changes in muscle growth factors that are associated with increases in muscle mass and strength in elderly hip fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in HSC protocol #97-0695 "Rehabilitation Intensification Post Hip Fracture"
* Community-dwelling
* Hip fracture within 16 weeks of the screening assessment for protocol 97-0695
* Persistent mobility and/or ADL impairments, but independent in ambulation
* Modified Physical Performance Test (PPT) score between 12 and 28

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134